CLINICAL TRIAL: NCT00002601
Title: High-Dose Doxorubicin and Ifosfamide Followed by Melphalan and Cisplatin for Patients With High-Risk and Recurrent Sarcoma
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94072; P30CA033572 (NIH); CHNMC-IRB-94072 (Registry Identifier: NCI PDQ); NCI-V94-0545; CDR0000063845 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Sarcoma
Keywords: metastatic osteosarcoma; recurrent childhood rhabdomyosarcoma; recurrent adult soft tissue sarcoma; recurrent osteosarcoma; adult rhabdomyosarcoma; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; previously treated childhood rhabdomyosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Filgrastim; Cisplatin; Doxorubicin; Ifosfamide; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin/Ifosfamide + Melphalan/CDDP + PSCT (Experimental): Cycle 1 Day -8 through Day -4 (96h) Doxorubicin 150 mg/m2 (CI) + Ifosfamide 14 g/m2 mixed with mesna (CI) Day -3 Mesna 3.5 g/m2 over 24 h Day -2 12.5% of stem cell reinfused.
  Cycle2 Day -11 Melphalan 75 mg/m2 + Cisplatin 100 mg/m2 Day -10 thru Day -6 G-CSF 5ug/kg Day -4 Melphalan 75 mg/m2 + Cisplatin 100 mg/m2 Day -3 12.5% if stem cell reinfused Day 0 37.5% of stem cell reinfused
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: melphalan; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim — 5 ug/kg daily following stem cell reinfusion
Drug: cisplatin — Course 2 - 100 mg/m2 at an infusion rate of 25 mg/hr
Drug: doxorubicin hydrochloride — Course 1 - 150 mg/m2 by continuous intravenous infusion for 96 hours.
Drug: ifosfamide — Course 1 - 14 gm/M2 by continuous intravenous infusion for 96 hours.
Drug: melphalan — Course 2 - 75 mg/m2 infused at a rate of 5 mg/minute
Procedure: peripheral blood stem cell transplantation — Administered on Day 0 following high-dose chemotherapy in both courses 1 and 2

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose combination chemotherapy and peripheral stem cell transplantation in treating patients who have advanced or recurrent sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of sequential high-dose chemotherapy with ifosfamide and doxorubicin followed by melphalan and cisplatin, each followed by autologous peripheral blood stem cell support, in patients with high-risk or advanced sarcomas. II. Determine the toxic effects of this regimen in these patients. III. Determine response rate and disease-free and overall survival in these patients treated with this regimen.

OUTLINE: Beginning at least 4 weeks prior to the start of chemotherapy, patients receive filgrastim (G-CSF) subcutaneously daily until the completion of peripheral blood stem cell (PBSC) harvesting. Beginning 5 days after the start of G-CSF, PBSCs are collected over several days. Patients who do not mobilize sufficient cells undergo bone marrow harvest. Regimen A: Patients receive high-dose ifosfamide IV and doxorubicin IV continuously over 96 hours on days -8 to -4. 12.5% of PBSCs or bone marrow are reinfused on day -2 and 37.5% are reinfused on day 0. Patients receive G-CSF IV beginning on day 0 and continuing until blood counts recover. Regimen B: Beginning at least 4 weeks after day 1 of Regimen A, patients receive high-dose melphalan IV followed immediately by cisplatin IV on days -11 and -4. Patients receive G-CSF IV on days -10 to -6. 12.5% of PBSCs or bone marrow are reinfused on day -3 and the remaining 37.5% are reinfused on day 0. Patients receive G-CSF IV beginning on day 0 and continuing until blood counts recover. Patients are followed monthly for 1 year, every 3 months for 1 year, and then as needed for 3 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed sarcomas in the following categories: Soft tissue sarcoma (STS) High-grade STS of the extremities Primary extending to fascia or locally recurrent At least 10 cm in greatest dimension or multifocal on surgical pathology Primary site controlled by surgery and/or radiotherapy High-grade truncal or head and neck sarcoma At least 10 cm in greatest dimension or any size with no surgical options for clear margins Primary site controlled by surgery and/or radiotherapy Locally recurrent disease in CR or PR after surgery, chemotherapy, or radiotherapy Metastatic STS in CR or PR after surgery, chemotherapy, or radiotherapy Osteosarcoma (OS) Extremity OS after neoadjuvant chemotherapy and surgical resection provided: Less than 50% necrosis in the surgical specimen LDH or alkaline phosphatase greater than 2 times normal at presentation Axial OS in CR or PR after chemotherapy and/or surgery Primary or recurrent metastatic OS in CR or PR after chemotherapy, surgery, and/or radiotherapy Ewing's sarcoma or primitive neuroectodermal tumor Primary site in CR or PR after chemotherapy, radiotherapy, or surgery Rib, pelvic, or axial skeleton primary Bulky tumor (at least 10 cm in greatest diameter) Primary or recurrent metastatic disease in CR or PR after surgery, chemotherapy, or radiotherapy Rhabdomyosarcoma Gross residual disease after primary treatment with surgery, chemotherapy, and radiotherapy Primary group IV or recurrent metastatic disease in CR or PR after chemotherapy and radiotherapy with or without surgery No brain metastasis No histologically confirmed bone marrow metastasis Prior metastases allowed with clearing of bone marrow at entry No contraindication to collection of mobilized stem cells or, if needed, autologous bone marrow

PATIENT CHARACTERISTICS: Age: 10 to 55 Performance status: Karnofsky 80-100% Hematopoietic: Absolute neutrophil count greater than 2,000/mm3 Platelet count greater than 150,000/mm3 Hemoglobin greater than 10 g/dL Hepatic: See Disease Characteristics Bilirubin less than 1.5 mg/dL AST and ALT less than 3 times normal Hepatitis B surface antigen negative Negative hepatitis C antigen test required in patients with hepatitis C antibody Renal: Creatinine less than 1.4 mg/dL Creatinine clearance greater than 75 mL/min Cardiovascular: LVEF at least 55% by MUGA or echocardiogram No history of significant cardiac disease Pulmonary: FEV1 greater than 2 liters PaO2 greater than 70 mm Hg on room air PaCO2 less than 42 mm Hg on room air DLCO greater than 60% predicted Other: No hearing loss of greater than 40 decibels HIV negative No organic or psychiatric CNS dysfunction that would preclude study No other medical or psychosocial problems that would place patient at unacceptable risk No history of other malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: More than 2 weeks since treatment to control primary or recurrent tumor Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No more than 2 prior chemotherapy regimens (including adjuvant therapy) Prior cumulative cisplatin dose less than 400 mg/m2 Prior cumulative doxorubicin dose less than 240 mg/m2 Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy to more than 20% of the bone marrow-containing axial skeleton No prior radiotherapy to the left chest wall Surgery: See Disease Characteristics

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 1994-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (1):
- Cancer Center and Beckman Research Institute, City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxorubicin/Ifosfamide + Melphalan/CDDP + PSCT
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Doxorubicin/Ifosfamide + Melphalan/CDDP + PSCT
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 31 [21 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 Bilirubin
Description: Criteria for early termination of this feasibility study: > 2 patients experience grade 4 or 5 hematologic toxicity or more that 3 patients experience grade 3 hematologic toxicity; > 2 patients experience grade 3 hepatic or gastrointestinal toxicity or > 3 patients are unable to receive the second cycle of treatment; > 2 patients experience grade 5 toxicity related to treatment regimen.
Time Frame: 2 years after completion of treatment
Measure: Number; unit: participants with Grade 3 Bilirubin
Arm/Group | Doxorubicin/Ifosfamide + Melphalan/CDDP + PSCT
Number analyzed (Participants) | 13
participants with Grade 3 Bilirubin | 3

2. Primary Outcome: Toxicities Counts
Description: Number of patients with grade 3 and 4 toxicities observed during cycles 1 & 2 using the Common Toxicity Criteria Version for Chemotherapy.
Time Frame: 2 months after completion of second cycle of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cycle 1: Day -8 through Day -4 (96h) Doxorubicin 150 mg/m2 (CI) + Ifosfamide 14 g/m2 mixed with mesna (CI) Day -3 Mesna 3.5 g/m2 over 24 h Day -2 12.5% of stem cell reinfused.
- Cycle 2: Day -11 Melphalan 75 mg/m2 + Cisplatin 100 mg/m2 Day -10 thru Day -6 G-CSF 5ug/kg Day -4 Melphalan 75 mg/m2 + Cisplatin 100 mg/m2 Day -3 12.5% if stem cell reinfused Day 0 37.5% of stem cell reinfused
Arm/Group | Cycle 1 | Cycle 2
Number analyzed (Participants) | 13 | 13
Participants
  Anemia | 8 | 3
  Leukopenia | 13 | 11
  Neutropenia | 13 | 11
  Febrile neutropenia | 13 | 9
  Thrombocytopenia | 13 | 11
  Mucositis | 13 | 1
  Bacteremia/sepsis | 2 | 4
  Hyperglycemia | 5 | 1
  Pulmonary function impairment (FEV1) | 1 | 0
  Pulmonary infiltrates | 0 | 2
  Diarrhea | 1 | 0
  Arrhythmia | 1 | 1
  Hematuria | 1 | 0
  Mood | 1 | 1
  Elevated PTT | 1 | 0

3. Secondary Outcome: 5-year Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 25% increase in the sum of the longest diameter of target lesions, or the appearance of new lesions.
Time Frame: Until disease progression, up to 5 Years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxorubicin/Ifosfamide + Melphalan/CDDP + PSCT
Number analyzed (Participants) | 13
percentage of participants | 23 [0 to 46]

4. Secondary Outcome: 5-year Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until death from any cause, up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxorubicin/Ifosfamide + Melphalan/CDDP + PSCT
Number analyzed (Participants) | 13
percentage of participants | 31 [14 to 70]

ADVERSE EVENTS:
Time Frame: Adverse events collected over a period of 45 months
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Doxorubicin/Ifosfamide + Melphalan/CDDP + PSCT
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin/Ifosfamide + Melphalan/CDDP + PSCT (N=13)
Dysrhythmias (Cardiac disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Partial Thromboplastin Time (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin/Ifosfamide + Melphalan/CDDP + PSCT (N=13)
Cerebellar (Nervous system disorders) | 9 (16)
Clinical (Physical Exam) (General disorders) | 9 (12)
Dysrhythmias (Cardiac disorders) | 6 (8)
Fluid Retention (Renal and urinary disorders) | 12 (20)
Hemorrhage (General disorders) | 12 (21)
Infection (Infections and infestations) | 12 (21)
Ischemia (Vascular disorders) | 7 (10)
Other Misc (General disorders) | 9 (31)
Pericardial (Cardiac disorders) | 7 (10)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 11 (18)
Stomatitis (General disorders) | 12 (22)
Weight (Food Intake) (Metabolism and nutrition disorders) | 8 (12)
Clinical Coagulation (Blood and lymphatic system disorders) | 9 (13)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
EF/CHF (Cardiac disorders) | 6 (9)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Hearing (Ear and labyrinth disorders) | 9 (16)
Eye disorder (Eye disorders) | 1 (1)
Vision (Eye disorders) | 9 (16)
Constipation (Gastrointestinal disorders) | 12 (21)
Diarrhea (Gastrointestinal disorders) | 13 (22)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (23)
Vomiting (Gastrointestinal disorders) | 13 (22)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (10)
Fever (no infection) (General disorders) | 11 (18)
Allergy (Immune system disorders) | 12 (21)
AGC (Investigations) | 12 (22)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline Phosphatase (Investigations) | 9 (12)
Amylase (Investigations) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Bilirubin (Investigations) | 9 (12)
Creatinine (Investigations) | 7 (8)
Creatinine increased (Investigations) | 1 (1)
Fibrinogen (Investigations) | 2 (3)
Hyperbilirubinemia (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Partial Thromboplastin Time (Investigations) | 7 (11)
Platelet count decreased (Investigations) | 1 (2)
Platelets (Investigations) | 12 (22)
Prothrombin Time (Investigations) | 9 (13)
SGOT/SGT (Investigations) | 9 (12)
WBC (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 12 (21)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (23)
Hypocalcemia (Metabolism and nutrition disorders) | 13 (23)
Hypoglycemia (Metabolism and nutrition disorders) | 12 (21)
Hypomagnesemia (Metabolism and nutrition disorders) | 13 (23)
Cortical/State of Consciousness (Nervous system disorders) | 9 (16)
Dizziness (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 10 (18)
Motor Activity (Nervous system disorders) | 9 (16)
Peripheral Nervous System Sensory (Nervous system disorders) | 9 (16)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Ideation (Psychiatric disorders) | 7 (12)
Insomnia (Psychiatric disorders) | 1 (1)
Mood (Psychiatric disorders) | 9 (16)
Hematuria (Renal and urinary disorders) | 7 (8)
Proteinuria (Renal and urinary disorders) | 7 (8)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (8)
Extensive Skin Rash (Skin and subcutaneous tissue disorders) | 8 (11)
Local Skin Rash (Skin and subcutaneous tissue disorders) | 8 (11)
Hypertension (Vascular disorders) | 2 (3)
Hypotension (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes